CLINICAL TRIAL: NCT00591890
Title: Phase IB Study to Evaluate the Biological Activity of Indibulin Using Positron-Emission Tomography (PET) Scans
Brief Title: Phase IB Study of Indibulin Using Positron-Emission Tomography (PET) Scans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBL1003
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — indibulin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: indibulin

INTERVENTIONS:
Drug: indibulin — dose escalation of indibulin given twice daily for 21 days, to be repeated every 28 days.
  Other Names: ZIO-301

SUMMARY:
Single arm, open label, Phase IB study of indibulin capsules in subjects with advanced solid tumors; eligible subjects will have a baseline PET scan showing a standardized uptake value (SUV) of ≥5.0 in ≥1 lesion on an 18F-FDG (fluorine-18-labeled deoxyglucose) scale.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of advanced cancer, refractory to standard therapies.
2. Received at least one prior therapy and requires additional treatment.
3. ≥18 years of age.
4. ECOG performance score ≤ 2 (see Appendix 3).
5. At least one measurable lesion as defined by RECIST (Response evaluation criteria in solid tumors) guidelines (see Appendix 4). If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions must NOT have been in a previously irradiated field or injected with biological agents.
6. PET scan showing a standardized uptake value (SUV) of ≥5.0 in at least 1 lesion on an 18F-FDG (fluorine-18-labeled deoxyglucose) scale.
7. Life expectancy ≥12 weeks.
8. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements, to be conducted <2 weeks prior to Day 1:

   * Creatinine ≤1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≥50 cc/minute
   * Total bilirubin ≤1.5 × ULN
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤2.5 × ULN
   * White blood cell count ≥3.0 × 109/L
   * Absolute neutrophil count (ANC) ≥1.5 × 109/L
   * Platelets ≥100 × 109/L
   * Hemoglobin ≥10 g/dL
9. Ability to tolerate repeated blood sampling and adequate vascular access.
10. Serum glucose levels ≤200 mg/dL.
11. Provide written informed consent in compliance with ZIOPHARM policies and the Independent Ethics Committee with jurisdiction over the site.
12. Subjects of childbearing potential must agree to use a barrier method of contraception throughout the study and for 3 months after study drug administration.

Exclusion Criteria:

1. New York Heart Association (NYHA) functional class ≥3 or myocardial infarction within 6 months (see Appendix 5).
2. Uncontrolled diabetes mellitus
3. Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation.
4. Pregnancy and/or lactation.
5. Uncontrolled systemic infection (documented with microbiological studies)
6. Any other anti-cancer or immunological therapy during the study or within 4 weeks of study entry. Mitomycin C or nitrosureas should not be given within 6 weeks of study entry.
7. Radiotherapy during the study or within 3 weeks of study entry.
8. Surgery within 4 weeks of start of study drug excluding tumor biopsy for pharmacodynamic parameters.
9. Investigational drug therapy outside of this trial during or within 4 weeks of study entry.
10. History of an invasive second primary malignancy diagnosed within the previous 3 years, except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
11. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
12. Any condition that is unstable or could jeopardize the safety of the subject and his/her compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
anti-tumor effect on PET Scan | 7 weeks

SECONDARY OUTCOMES:
toxicities | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, Study Director — Alaunos Therapeutics
Locations (1):
- Santa Monica, California, United States

REFERENCES:
- [Derived] Kapoor S, Srivastava S, Panda D. Indibulin dampens microtubule dynamics and produces synergistic antiproliferative effect with vinblastine in MCF-7 cells: Implications in cancer chemotherapy. Sci Rep. 2018 Aug 17;8(1):12363. doi: 10.1038/s41598-018-30376-y. PMID 30120268